CLINICAL TRIAL: NCT06334003
Title: Cardiometabolic Function in Offspring, Mother and Placenta After Assisted Reproductive Technology
Acronym: COMPART
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Anja Bisgaard Pinborg, Clinical Professor, Rigshospitalet, Denmark
Other Study IDs: H-23071266
Record Dates: First submitted 2024-02-26; First posted 2024-03-27 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: ART; IVF; Children, Only; Cardiovascular Disease Other
Keywords: Frozen embryo transfer; Cardiovascular; Metabolic; IVF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- FET-group: Children conceived by frozen embryo transfer
- Fresh ET-group: Children conceived by fresh embryo transfer
- NC group: Naturally conceived children

SUMMARY:
The overall objective is to establish the first-of-its-kind longitudinal cohort of pregnant women, biological fathers/partners and offspring from pregnancies achieved by frozen embryo transfer (FET), fresh-embryo transfer (fresh ET) and naturally conceived (NC) to investigate maternal cardiometabolic profiles, fetal growth patterns and placental function during pregnancy as well as metabolic and endocrine health in the offspring. Additionally, the aim is to explore genetic and epigenetic patterns in placenta, fetus and parents. As secondary objectives, the investigator group will examine telomere length and minipuberty hormones in children born after FET, fresh-ET and NC.

DETAILED DESCRIPTION:
Background and research gap: Increasing use of assisted reproductive technology (ART) necessitates vigilance on the health of the offspring. The use of frozen embryo transfer (FET) in ART increases the risk of the children being born large-for-gestational-age (LGA) compared to conventional fresh embryo transfer (fresh ET) and naturally conceived children (NC). In general, children born LGA are predisposed to childhood obesity and later metabolic syndrome, thus FET may increase the societal burden of this. The mechanism between FET and LGA is unclear and its impact on neonatal body composition and metabolic health is unknown.

Hypothesis and objectives: The growth hormone (GH) - insulin-like growth factor (IGF) axis plays an essential role in fetal growth and is also linked to metabolic disease due to its interactions with insulin. Thus, the investigator group hypothesize that FET imposes epigenetic alterations towards the GH-IGF-axis leading to enhanced fetal growth and a potential persisting phenotype of metabolic dysfunction. The objective is to determine the effect of endocrine growth factors, maternal metabolic profile, and placental function on intrauterine growth patterns as well as early postnatal body composition and metabolic profile in children born after ART with FET compared to children born after fresh ET and NC children.

Methods and outcomes: The investigator group will conduct a prospective cohort study including women pregnant by FET (N=200), fresh ET (N=200) and NC children (N=200). The women will undergo three examinations during pregnancy with blood sampling (analyzed for GH-IGF-related growth factors and metabolic biomarkers), fetal biometry and doppler ultrasound. For a subpopulation the placenta will be collected at delivery. The expression of placental growth factors will be determined using western blot and qPCR and epigenetic alterations assessed by DNA methylation using targeted CpG arrays. The newborns will be examined within two weeks of birth with blood samples (analyzed for growth factors, glucose-metabolism markers, lipids, and cytokines) and a DEXA-scan to evaluate body composition. Information on ART-procedure, obstetric adverse events, birth weight and neonatal complications will be available from electronic health records. The outcomes are grouped in three work packages comparing the differences between FET, fresh ET, and NC in 1) maternal growth factors and metabolic profile and the relationship with fetal growth trajectories, 2) expression and DNA methylation of GH-IGF-axis components in placental tissue, 3) body composition, metabolic profile and DNA methylation of regions related to the GH-IGF axis in neonates.

Significance: It is crucial to understand the mechanism between FET and LGA and its impact on metabolic health in children in order to determine the safest ART technique. The investigator group expect that the results will identify the role of the GH-IGF axis in the pathogenesis of FET-induced LGA and its associated metabolic risk which may highlight potential biomarkers of abnormal fetal growth and therapeutic targets for prevention of obesity and metabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women who have either had fertility treatment at Rigshospitalet or Herlev Hospital (FET and fresh ET groups) or are scheduled for prenatal ultrasounds at Rigshospitalet or Herlev Hospital (NC group) will be screened for eligibility. Inclusion must happen before their routine ultrasound scan in 1. trimester.

Exclusion Criteria:

* Maternal pregestational diabetes type 1 or 2
* Non-singleton pregnancies
* Maternal pregestational BMI > 35 kg/m2
* Severe maternal co-morbidity
* Oocyte donation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be recruited from the Capital Region of Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Offspring body composition | Assessed at 2,5 months of age
  Total fat mass (in gram) assessed by air displacement plethysmography (PEA POD).
Maternal cardiometabolic profile | One times during each trimester
  Fetal growth patterns determined by ultrasound

SECONDARY OUTCOMES:
Epigenetic in placenta and cord blood | 2 years
  Differences between ovulatory FET, programmed FET, fresh ET and NC
Early markers of reproductive function in FET, fresh-ET and NC children: LH, FSH, SHBG, AMH, androgens, estrogens (SDS) | 3 years
  Bloodsamples: Differences between ovulatory FET, programmed FET, fresh ET and NC
Telomere length in children born after FET, fresh-ET and NC children | 3 years
  Differences between ovulatory FET, programmed FET, fresh ET and NC in 1) LTL in newborns and 2) parental LTL

CONTACTS AND LOCATIONS:
Overall Officials: Anja B. Pinborg, Prof., MD, Principal Investigator — Fertility Department, Rigshospitalet; Rikke B. Jensen, MD, Ass. prof, Study Chair — Dept. of Paediatric and Adolescent Medicine, Herlev Hospital
Locations (3):
- Denmark (3):
  - Fertility Clinic, Rigshospitalet, Copenhagen University Hospital, Copenhagen
  - Department of Fetalmedicin, Herlev Hospital, Copenhagen
  - Dept. of Paediatric and Adolescent Medicine, Herlev Hospital, Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kjaer ASL, Vestager ML, Blixenkrone-Moller E, Asserhoj LL, Kloppenborg JT, Lossl K, Ekelund CK, Rode L, Hjort L, Hoffmann ER, Lyng Forman J, Beck Jensen R, Pinborg A. Cardiometabolic function in Offspring, Mother and Placenta after Assisted Reproductive Technology (COMPART): a prospective cohort study. BMJ Open. 2025 Sep 16;15(9):e105754. doi: 10.1136/bmjopen-2025-105754. PMID 40957860